CLINICAL TRIAL: NCT01403324
Title: Comparison of Dosimetry Following Preparation With Either rhTSH or After Withdrawal of Thyroid Hormone Suppression Therapy in Patients With Metastatic or Locally Advanced Differentiated Thyroid Cancer
Brief Title: Comparison of Dosimetry After rhTSH or Withdrawal of Thyroid Hormone in Metastatic or Locally Advanced Thyroid Cancer
Acronym: DOSIMETA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DOSIMETA IGR2010/1645
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Thyroid Cancer; Metastases
Keywords: metastatic or locally advanced differentiated thyroid cancer; planned for a therapeutic activity of 131I after thyroid hormone withdrawal
MeSH Terms: conditions — Thyroid Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TSH stimulation (Other): rh TSH stimulation followed by thyroid hormon withdrawal
  Interventions: Drug: TSH stimulation

INTERVENTIONS:
Drug: TSH stimulation — rh TSH stimulation followed by thyroid hormon withdrawal

SUMMARY:
Metastases of thyroid cancer with iodine uptake are treated with repeated activity of I-131 administered after thyroid hormone withdrawal. The goal of thyroid hormone withdrawal is to treat patients with elevated thyrotropin stimulated hormone (TSH), a hormone secreted by the pituitary, a gland just located under the brain. Another way to obtain elevated TSH levels is to perform intramuscular injection of recombinant human TSH, a hormone produced pharmaceutically. The goal of this study is to know whether the radioiodine uptake by the metastases is similar after rhTSH administration or after thyroid hormone withdrawal.

DETAILED DESCRIPTION:
Patients will undergo a rhTSH stimulation, staying on thyroid hormone treatment. Following 2 administration of rhTSH an injection of I-124 will be performed. Positron emission tomography with computed tomography scans (PET/CT), blood tests, and measurements of whole body radioactivity will occurred during the 4 to 96 hours following I-124 administration in order to perform dosimetry (i.e.) to estimate the radiation dose delivered to the metastases. After 4 weeks under thyroid hormones patients will undergo thyroid hormone withdrawal and a new administration of I-124 will be performed. The same dosimetry study will be realized with PET/CT, blood tests, and measurements of whole body radioactivity. A therapeutic activity of I-131will then be administered followed by whole body scan realized 24 to 72 hours after the administration of I-131. Dosimetry studies will be compared in order to determine whether rhTSH stimulation can replace thyroid hormone withdrawal for the treatment of distant metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with thyroid cancer and known measurable (>1cm) distant metastases demonstrating radioiodine uptake on a previous whole body scan
2. Patients planned for a therapeutic activity of 131I after thyroid hormone withdrawal
3. Age >18 years
4. Previous treatment with radioiodine more than 6 months before inclusion.
5. Serum TSH level <0.5 mU/L
6. Normal renal function with a creatinine clearance estimation using the Cockcroft-Gault formula > 60 ml/ml
7. Effective means of contraception for female patient, at risk of pregnancy
8. Written informed consent

Exclusion Criteria:

1. Patients whose majority of tumoral lesions disclose FDG uptake without radioactive iodine uptake
2. Iodine excess (< 50 μg/dl)
3. Large or diffuse bone or brain metastases
4. Patients with multiple small tumor foci less than 1 cm in diameter, such as miliary spread to the lungs
5. Patients already included in a therapeutic trial with an experimental medicine
6. Pregnancy and breast feeding patients
7. Subject with any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures
8. Treatment with antivitamin k

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
the 124 I uptake after TSH stimulation | 4 to 96 hours
  For each patient, the 124 I uptake after TSH stimulation (a marker of radiation absorbed dose) will be compared to the uptake after thyroid withdrawal in all lesions (up to 16 lesions per patient maximum). A decrease in the residence time of more than 2.5 fold in 25% or more of the lesions is considered unacceptable.

SECONDARY OUTCOMES:
The activity of 131I that should be administered according to each TSH stimulation method | 96 hours
  To determine the activity of 131I that should be administered following rhTSH to deliver a radiation absorbed dose similar to that delivered under hypothyroid conditions. A calculated activity above 250mCi is considered unacceptable.
Radiation exposure of the blood | 4 to 96 hours
  The radiation exposure of the blood, calculated from blood samples and whole body radioactivity measurements

CONTACTS AND LOCATIONS:
Overall Officials: Sophie LEBOULLEUX, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France